CLINICAL TRIAL: NCT06576115
Title: Treatment of Patients With Metastatic Pancreatic Cancer With Gemcitabine and Nab-Paclitaxel and Amplitude-Modulated Radiofrequency Electromagnetic Fields (AM RF EMF)
Brief Title: Gemcitabine, Nab-paclitaxel Plus the TheraBionic P1 (an Amplitude-Modulated Radiofrequency Electromagnetic Fields) Device to Treat Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Associate Center Director, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-104
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Gemcitabine/Nab-Paclitaxel plus TheraBionic Device (Experimental): Metastatic pancreatic cancer patients will be treated with amplitude-modulated radiofrequency electromagnetic fields using TheraBionic device in combination with standard chemotherapy, gemcitabine- nab-paclitaxel. amplitude-modulated radiofrequency electromagnetic fields will be delivered by the TheraBionic device.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Device: TheraBionic P1

INTERVENTIONS:
Drug: Nab paclitaxel — 125 mg/m2 weekly, on days 1,8, and 15 or on days 1 and 15 as a 30-40 minute infusion administered first
  Other Names: Abraxane
Drug: Gemcitabine — 1000 mg/m2 weekly, on day 1,8 and 15 or 1000 mg/m2 weekly, on day 1 and 15 over 30 minutes after nab- paclitaxel infusion
  Other Names: Gemzar
Device: TheraBionic P1 — This treatment consists of delivering preset low levels of radio waves into the body with a spoon-shaped antenna placed in the mouth, three times a day, for an hour each time.

SUMMARY:
The goal of this study is to learn if the combination of nab-paclitaxel, gemcitabine and an Amplitude-Modulated Radiofrequency Electromagnetic Fields device (Therabionic P1) is safe and effective for patients with adenocarcinoma of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven advanced metastatic adenocarcinoma of the pancreas. Patients with mixed tumor with predominant adenocarcinoma pathology can be enrolled.
* One or more measurable metastatic tumors per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) on imaging studies CT or MRI or PET scans
* If female patient is of childbearing potential must have a negative serum pregnancy test (βhCG) documented up to 48 hrs prior to administration of chemotherapy.
* Females of childbearing potential and males with female partners of childbearing potential, if sexually active, must agree to use two forms of contraception during the period of administration of study drug and up to 6 months after the end of treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Age above 18 years
* Based on prior studies, patients 80 years of age and older are considered to be at higher risk for fatal neutropenic sepsis. These patients should be thoroughly evaluated including geriatric assessment prior to enrollment. Clinical judgment should be exercised regarding patients' susceptibility for sepsis or infection (presence of biliary tract infection, uncontrolled diabetes, etc.). The patients in this age group should be not enrolled should there be any concern for rapid deterioration of clinical and functional status.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Parameter Levels:

Absolute neutrophil count (ANC) ≥ 1,500/mcL Platelets > 100,000/mcL Total bilirubin ≤ 1.5 X institutional upper limit of normal AST(SGOT)/ALT(SGPT) < 2.5 X ins Creatinine ≤ 1.5 X institutional upper limit of normal Or CrCL > 50

* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Patients who have had chemotherapy with gemcitabine and/or nab-paclitaxel within six months prior to entering the study in the adjuvant or neo-adjuvant setting.
* Patients receiving any other investigational agents.
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine and nab-paclitaxel.
* No history of malignancy in last 3 years except cervical cancer in situ, adequately treated basal cell or squamous cell carcinoma of skin or treated low risk prostate cancer, who are considered to be eligible.
* Patients receiving calcium channel blockers and any agent blocking L-type of T-type Voltage Gated Calcium Channels such as amlodipine, nifedipine, ethosuximide are not allowed in the study unless their medical treatment is modified to exclude calcium channel blockers prior to enrollment. (Refer to Appendix D for a comprehensive list of excluded medications)
* Patients with active and uncontrolled bacterial, viral or fungal infection requiring systemic therapy. Patients can be reevaluated for the study if the infection is deemed to be under control and the systemic therapy is completed.
* Uncontrolled intercurrent illness including, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or could compromise patients' safety.
* Patient with known diagnosis of interstitial lung disease, sarcoidosis, pulmonary fibrosis or pneumonitis.
* Pregnant women are excluded from this study because of potential risk for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy and AM RF EMF, patients who are breastfeeding will be excluded to participate in this study.
* Patient has localized resectable or locally advanced tumor.
* Patients has undergone major surgery, other than diagnostic surgery or procedures, within 4 weeks prior to the treatment day.
* Patients is unable to comply with study procedures or anticipating a situation that would result in a treatment break for 14 or more consecutive days after the start of the study.
* Patient is enrolled in any other clinical interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
6 Month Progression-Free Survival Rate (PFS 6) | 6 months
  Progression-free survival (PFS) is defined from the time of study treatment initiation until progression or death of any cause, whichever occurs first. The six months PFS rate (PFS 6) is defined as the proportion of patients alive and progression-free at six months from treatment initiation. PFS will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines.

SECONDARY OUTCOMES:
Adverse Event Incidence | Up to 1 year
  Evaluate the safety and tolerability of the combination of nab-paclitaxel, gemcitabine and AM RF EMF categorized and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5). The adverse event incidence rate will be defined as a proportion of patients who experience adverse events among the safety population.
Median Progression Free Survival (PFS) | Up to 1 year
  PFS is defined from the time of study treatment initiation until progression or death of any cause, whichever occurs first. PFS will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines. The median PFS will be estimated using Kaplan-Meier estimate.
6-month Overall Status rate (OS 6) | 6 Months
  Overall survival (OS) is defined from the time of study treatment initiation until the death of any cause. The six months OS rate (OS 6) is defined as the proportion of patients alive at six months from treatment initiation.
Median OS | Up to 1 year
  OS is defined from the time of study treatment initiation until death of any cause. The median OS will be estimated using Kaplan-Meier estimate.
Objective Response Rate (ORR) | Up to 1 year
  ORR is defined as the proportion of patients with partial or complete responses based on Radiographic Determination of Treatment Response by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) by CT Scan or MRI:
  1. Complete Response (CR): Complete disappearance of all target and non-target lesions (with the exception of lymph nodes mentioned below). No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline.
  2. Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions.
Disease Control Rate (DCR) | Up to 1 year
  Disease control rate is defined as the proportion of patients with disease control (complete or partial response or stable disease) based on RECISTv1.1 criteria:
  1. Complete Response (CR): Complete disappearance of all target and non-target lesions (with the exception of lymph nodes mentioned below). No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline.
  2. Partial Response (PR): Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions.
  3. Stable disease: Does not qualify for CR, PR, Progression or Symptomatic Deterioration. All target measurable lesions must be assessed using the same techniques as baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Shields, M.D. PhD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (7):
- United States (7):
  - Karmanos Cancer Institute at McLaren Clarkston, Clarkston, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at McLaren Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Karmanos Cancer Institute at McLaren Lapeer Region, Lapeer, Michigan
  - Karmanos Cancer Institute at McLaren Northern Michigan, Petoskey, Petoskey, Michigan
  - Karmanos Cancer Institute at McLaren Port Huron, Port Huron, Michigan